CLINICAL TRIAL: NCT00198900
Title: Use of Modified Foods in the Dietary Treatment of Type II Diabetes Mellitus: Knowledge Assessment
Brief Title: Diabetes Knowledge Assessment
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: American Diabetes Association (Other)
Other Study IDs: ADA2000-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2000-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: survey of information

SUMMARY:
To assess the knowledge of both type 2 diabetics and non-diabetics on diabetes, nutrition, and exercise. Although type 2 diabetics should know more about their disease and its needs, it is not expected they will know significantly more than the lay public.

DETAILED DESCRIPTION:
A validated survey about diabetes, nutrition, obesity, and exercise will be dispersed to type 2 diabetics and non-diabetics, and then analyzed.

ELIGIBILITY:
Inclusion Criteria:

type 2 diabetic or non-diabetic, age 18 and over

Exclusion Criteria:

type 1 diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2000-01; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Lutherville, Maryland, United States